CLINICAL TRIAL: NCT02365896
Title: Comparison of Short Term Outcomes Between Totally Laparoscopic and Laparoscopy-Assisted Distal Gastrectomy With Billroth-II Reconstruction and D2 Lymphadenectomy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLDG vs. LADG
Record Dates: First submitted 2015-01-23; First posted 2015-02-19 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-01

CONDITIONS: Total Laparoscopic Distal Gastrectomy; Locally Advanced Gastric Cancer

ARMS (1):
- TLDG or LADG (Other): To complete the distal gastrectomy with Billroth-II reconstruction and D2 lymphadenectomy for locally advanced gastric cancer with TLDG or LADG
  Interventions: Procedure: TLDG or LADG

INTERVENTIONS:
Procedure: TLDG or LADG

SUMMARY:
Prospective Randomized Controlled Multicenter Clinical Trial for Comparison of Safety Between Totally Laparoscopic Distal Gastrectomy(TLDG) and Laparoscopy-Assisted Distal Gastrectomy(LADG) With Billroth-II Reconstruction and D2 Lymphadenectomy for Locally Advanced Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of gastric cancer was confirmed by pathological examination
* Preoperative staging as cT2-4aN0-3M0 according to AJCC-7th
* No accompany with another cancer
* ECOG 0-1
* ASA I-III
* Agreement

Exclusion Criteria:

* Pregnant or suckling period
* Patients with a history of preoperative chemoradiotherapy
* Patients with unable to finish D2 lymphadenectomy or R0 resection
* Laparoscopic surgery contraindications
* Serious organ disfunction
* Accompany with serious mental disease
* Continuous treatment with steroid in 1 month
* Disagreement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
postoperative early anastomotic morbidity | 30 days

SECONDARY OUTCOMES:
Flatus time | 7 days
Quality of life | 30 days
  estimated with EORTC QLQ-C30V3、EORTC QLQ-STO22
Postoperative hospital stay | 30 days
Pain score | 10 days
Postoperative inflammation response | 10 days
  using C-reactive protein、IL-6、WBC and so on postoperative 1,3,5,7 days
Nutrition | 30 days
  NRS-2002 and PG-SGA in 30 days

REFERENCES:
- [Background] Ikeda O, Sakaguchi Y, Aoki Y, Harimoto N, Taomoto J, Masuda T, Ohga T, Adachi E, Toh Y, Okamura T, Baba H. Advantages of totally laparoscopic distal gastrectomy over laparoscopically assisted distal gastrectomy for gastric cancer. Surg Endosc. 2009 Oct;23(10):2374-9. doi: 10.1007/s00464-009-0360-3. Epub 2009 Mar 5. PMID 19263143
- [Background] Han G, Park JY, Kim YJ. Comparison of short-term postoperative outcomes in totally laparoscopic distal gastrectomy versus laparoscopy-assisted distal gastrectomy. J Gastric Cancer. 2014 Jun;14(2):105-10. doi: 10.5230/jgc.2014.14.2.105. Epub 2014 Jun 30. PMID 25061537
- [Background] Oki E, Sakaguchi Y, Ohgaki K, Saeki H, Chinen Y, Minami K, Sakamoto Y, Toh Y, Kusumoto T, Maehara Y. Feasibility of delta-shaped anastomoses in totally laparoscopic distal gastrectomy. Eur Surg Res. 2011;47(4):205-10. doi: 10.1159/000332850. Epub 2011 Oct 13. PMID 22004901
- [Background] Kim BS, Yook JH, Choi YB, Kim KC, Kim MG, Kim TH, Kawada H, Kim BS. Comparison of early outcomes of intracorporeal and extracorporeal gastroduodenostomy after laparoscopic distal gastrectomy for gastric cancer. J Laparoendosc Adv Surg Tech A. 2011 Jun;21(5):387-91. doi: 10.1089/lap.2010.0515. Epub 2011 May 11. PMID 21561328
- [Background] Kim MG, Kim KC, Kim BS, Kim TH, Kim HS, Yook JH, Kim BS. A totally laparoscopic distal gastrectomy can be an effective way of performing laparoscopic gastrectomy in obese patients (body mass index>/=30). World J Surg. 2011 Jun;35(6):1327-32. doi: 10.1007/s00268-011-1034-6. PMID 21424875
- [Background] Lee J, Kim D, Kim W. Comparison of laparoscopy-assisted and totally laparoscopic Billroth-II distal gastrectomy for gastric cancer. J Korean Surg Soc. 2012 Mar;82(3):135-42. doi: 10.4174/jkss.2012.82.3.135. Epub 2012 Feb 27. PMID 22403746
- [Background] Woo J, Lee JH, Shim KN, Jung HK, Lee HM, Lee HK. Does the Difference of Invasiveness between Totally Laparoscopic Distal Gastrectomy and Laparoscopy-Assisted Distal Gastrectomy Lead to a Difference in Early Surgical Outcomes? A Prospective Randomized Trial. Ann Surg Oncol. 2015;22(6):1836-43. doi: 10.1245/s10434-014-4229-x. Epub 2014 Nov 14. PMID 25395149
- [Background] Song KY, Park CH, Kang HC, Kim JJ, Park SM, Jun KH, Chin HM, Hur H. Is totally laparoscopic gastrectomy less invasive than laparoscopy-assisted gastrectomy?: prospective, multicenter study. J Gastrointest Surg. 2008 Jun;12(6):1015-21. doi: 10.1007/s11605-008-0484-0. Epub 2008 Feb 7. PMID 18256884